CLINICAL TRIAL: NCT04281108
Title: Fluticasone Propionate Oral Dispersible Tablet Formulation in Eosinophilic Esophagitis: A Two-Part, Randomized, Double-blind, Placebo-Controlled Study of APT-1011 With an Open-label Extension, in Adult Subjects With Eosinophilic Esophagitis
Brief Title: Efficacy and Safety APT-1011 in Adult Subjects With Eosinophilic Esophagitis (EoE) (FLUTE-2)
Acronym: FLUTE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ellodi Pharmaceuticals, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-1011-003
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Eosinophilic Esophagitis
Keywords: APT-1011; Esophagitis; Eosinophilic Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Fluticasone; Anti-Inflammatory Agents; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Anti-Asthmatic Agents; Respiratory System Agents; Anti-Allergic Agents
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — APT-1011; Fluticasone; Endoscopy, Digestive System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APT-1011 (Experimental): APT-1011 3 mg HS
  Interventions: Drug: APT-1011; Procedure: Esophagogastroduodenoscopy
- Placebo (Placebo Comparator): HS
  Interventions: Drug: Placebo oral tablet; Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Drug: APT-1011 — APT-1011 is an orally disintegrating tablet that includes fluticasone propionate as its active ingredient.
  Other Names: fluticasone propionate
  Arms: APT-1011
Drug: Placebo oral tablet — Placebo orally disintegrating tablet.
  Other Names: PBO
  Arms: Placebo
Procedure: Esophagogastroduodenoscopy — Esophagogastroduodenoscopy (EGD) is a test that involves an endoscope, a lighted camera on the end of a tube, that is passed down a subject's throat to visualize their esophagus.

SUMMARY:
This is a 2-part randomized, double-blind, placebo-controlled study followed by an open-label extension (OLE) of APT-1011 in adults with EoE.

Part A will evaluate the efficacy and safety of APT-1011 3 mg administered hora somni (HS; at bedtime) for the induction of response to treatment (histologic and symptomatic) over 12 weeks.

Part B will evaluate histological relapse-free status in patients re-randomized to continue APT-1011 or placebo (active treatment withdrawal) until Week 52.

Part C, the OLE, will continue until regulatory approval of APT-1011 or Sponsor termination of the study.

DETAILED DESCRIPTION:
This is a 2-part randomized, double-blind, placebo-controlled study followed by an OLE of APT-1011 in adults with EoE.

Part A will evaluate the efficacy and safety of APT-1011 3 mg administered HS for the induction of response to treatment (histologic and symptomatic) over 12 weeks.

At Week 14, subjects will move into Part B. Subjects with histological response to APT-1011, defined as ≤6 peak eos/HPF, will be re-randomized to continue APT-1011 or receive placebo (active treatment withdrawal). APT-1011 histological non-responders will continue APT-1011, and placebo histological non-responders will receive APT-1011 3 mg HS. Placebo histological responders will continue placebo. The double-blind will be sustained throughout Part B. Histological responder status will be determined at the time of esophagogastroduodenoscopy (EGD) in Part B (at or prior to Week 52, depending on unscheduled EGDs performed when the Investigator deems the subject's symptoms necessitate EGD) and is defined as ≤6 peak eos/HPF.

At Week 52, subjects may enter Part C, an open-label single-arm extension phase, and continue study drug uninterrupted. Part C will terminate upon regulatory approval of APT-1011 or Sponsor termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of informed consent or assent
2. Each subject must read, understand, and provide consent on the ICF for this study and be willing and able to adhere to study-related treatment regimens, procedures, and visit schedule
3. Diagnosis or presumptive diagnosis of EoE that is confirmed during the Screening period by histology that demonstrates ≥15 peak eos/HPF. In order to ensure that a diagnosis can be made, at least 6 biopsies should be taken including both proximal and distal specimens (at least 3 each). Mid-esophageal biopsies are not required (optional). HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens (0.3 mm^2) and 22 mm ocular.

   1. Esophagogastroduodenoscopies and biopsies are to be obtained during the Screening period
   2. Biopsies will be read by a central pathologist
   3. Esophagogastroduodenoscopies and biopsies performed outside the study will not be accepted to meet eligibility criteria
   4. Optional biopsies may be taken and processed locally for local use, if specified in the local ICF. If serious pathology is unexpectedly encountered biopsies of such lesions must be processed locally
4. Have a subject-reported history of ≥6 episodes of dysphagia in the 14 days prior to baseline
5. Completion of the daily diary on at least 11 out of the 14 days during the 2-week Baseline Symptom Assessment

Exclusion Criteria:

1. Have known contraindication, hypersensitivity, or intolerance to corticosteroids
2. Have a contraindication to, or factors that substantially increase the risk of, EGD procedure or esophageal biopsy or have narrowing of the esophagus that precludes EGD with a standard 9 mm endoscope
3. Have history of an esophageal stricture requiring dilatation within the 12 weeks prior to Screening
4. Have any physical, mental, or social condition or history of illness or laboratory abnormality that in the Investigator's judgment might interfere with study procedures or the ability of the subject to adhere to and complete the study or increase the safety risk to the subject such as uncontrolled diabetes or hypertension
5. History or presence of oral or esophageal mucosal infection whilst using inhaled or nasal corticosteroids
6. Have any mouth or dental condition that prevents normal eating (excluding braces)
7. Have any condition affecting the esophageal mucosa or altering esophageal motility other than EoE, including erosive esophagitis (grade B or higher as per the Los Angeles Classification of Gastroesophageal Reflux Disease; hiatus hernia longer than 3 cm, Barrett's esophagus, and achalasia)
8. Use of systemic (oral or parenteral) corticosteroids within 60 days before Screening, use of swallowed corticosteroids within 30 days before Screening
9. Initiation of either inhaled or nasal corticosteroids or high-potency dermal topical corticosteroids within 30 days before Screening
10. Use of calcineurin inhibitors or purine analogues (azathioprine, 6-mercaptopurine) in the 12 weeks before Screening
11. Use of potent cytochrome P450 (CYP) 3A4 inhibitors (eg, ritonavir and ketoconazole) in the 12 weeks before Screening
12. Initiation of an elimination diet or elemental diet within 30 days before Screening (diet must remain stable after signing ICF)
13. Morning (07:00 to 09:00, or as close to that window as possible) serum cortisol level ≤5 μg/dL (138 nmol/L) that is not responsive to adrenocorticotropic hormone (ACTH) stimulation: defined as a serum cortisol level <16 μg/dL (440 nmol/L) at 60 minutes with ACTH stimulation test using 250 μg cosyntropin (i.e., an abnormal result on the ACTH stimulation test)
14. Use of biologic immunomodulators in the 24 weeks before Screening (allergy desensitization injection or oral therapy is allowed as long as the course of therapy is not altered during the study period)
15. Subjects who have initiated, discontinued, or changed dosage regimen of histamine H2 receptor antagonists, antacids or antihistamines for any condition such as gastro-esophageal reflux disease within 4 weeks before qualifying endoscopy during Screening. If already receiving these drugs, the dosage must remain constant throughout the study
16. Subjects who have changed dosage regimen of PPIs within 8 weeks before qualifying endoscopy. If already receiving PPIs, the dosage must remain constant throughout the study
17. Infection with hepatitis B, hepatitis C, or human immunodeficiency virus
18. Have gastrointestinal bleeding or documented active peptic ulcer within 4 weeks prior to Screening or entering a new study period
19. Have chronic infection such as prior or active tuberculosis, active chicken pox or measles or absence of prior measles, mumps and rubella vaccine. Subjects with tuberculosis exposure or who live in, or travel to, high endemic areas should be assessed locally for tuberculosis before consideration for the study
20. Immunosuppression or immunodeficiency disorder
21. Have a history or presence of Crohn's disease, celiac disease, or other inflammatory disease of the gastrointestinal tract, including eosinophilic gastroenteritis
22. Have current drug abuse in the opinion of the Investigator.
23. Have current alcohol abuse in the opinion of the Investigator.
24. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
25. Sexually active females of childbearing potential who do not agree to follow highly effective contraceptive methods through the End of Study visit
26. Have received an investigational product, as part of a clinical trial within 30 days (or 5 half-lives, whichever is longest) of Screening. Subjects who are currently participating in observational studies or enrolled in patient registries are allowed in this study
27. Have participated in a prior study with investigational product APT-1011

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Week 12 histologic responder rates | Week 12
  To compare the Week 12 histologic responder rates (≤ 6 peak eosinophils [eos]/high power field [HPF]) for APT-1011 3 mg HS with that for placebo. HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens (0.3 mm^2) and 22 mm ocular
Mean change in number of dysphagia episodes | Week 0 to Week 12
  To compare the mean change in number of dysphagia episodes from baseline to Week 12 for APT-1011 3 mg HS with that for placebo
Histologic responder rates at the end of the Randomized Withdrawal Phase (RWS) | Week 12 to Week 52
  To compare the histologic responder rates (≤ 6 peak eos/HPF) for APT-1011 responders randomized to continuing APT-1011 3 mg HS (maintenance) with responders randomized to placebo (withdrawal of APT-1011 3 mg HS) at the end of the RWS
Percentage subjects with complete symptomatic response at the end of the RWS | Week 0 to Week 52
  Percentage of subjects with complete symptomatic response (i.e., no dysphagia episodes for the 14 consecutive days prior to the end of the randomized withdrawal phase) at the end of the randomized withdrawal phase, in the RWS APT-1011 3 mg HS arm versus placebo arm

SECONDARY OUTCOMES:
Change in EREFs from Week 0 to Week 12 | Week 0 to Week 12
  To compare endoscopic appearance evaluated by the mean change from baseline to Week 12 in Eosinophilic Esophagitis Endoscopic Reference Score (EREFs) for APT-1011 3 mg HS with that for placebo.
Percentage of subjects with <1 peak eos/HPF at Week 12 | Week 12
  To compare the percentage of subjects with <1 peak eos/HPF at Week 12 for APT-1011 3 mg HS with that for placebo.
Mean change in PROSE Symptom Burden Score | Week 0 to Week 12
  To compare the mean change from baseline to Week 12 in the day-level symptom burden utilizing the Patient Reported Outcomes Symptoms of EoE (PROSE) for APT-1011 3 mg HS with that for placebo.
Mean Change in PROSE Day-Level Difficulty Swallowing | Week 0 to Week 12
  To compare the mean change from baseline to Week 12 in day-level difficulty swallowing using the Patient Reported Outcomes Symptoms of EoE (PROSE) for APT-1011 3 mg HS with that for placebo. Each symptom is rated on a numeric rating scale (NRS) with values ranging from 0 (not at all) to 10 (as bad as I can imagine).
Mean Histologic Change from Baseline to Week 12 | Week 0 to Week 12
  To compare mean histologic change from baseline to Week 12 for APT-1011 3 mg HS with that for placebo.
Percentage of Subjects with <15 peak eos/HPF | Week 12
  To compare the percentage of subjects with <15 peak eos/HPF for APT-1011 3 mg HS with that for placebo.
Mean Number of Dysphagia-free Days | Week 0 to Week 12
  To compare the mean number of dysphagia-free days from baseline to Week 12 for APT-1011 3 mg HS with that for placebo
Mean Change in Dysphagia Episodes | Week 0 to Week 52
  To compare mean change in number of dysphagia episodes from baseline to the end of RWS for APT-1011 responders randomized to continue APT-1011 3 mg HS with responders randomized to placebo (withdrawal of APT-1011 3 mg HS)
Mean Change in EREFs from Week 0 to Week 52 | Week 0 to Week 52
  To compare endoscopic appearance evaluated by the mean change from baseline to the end of RWS, in Eosinophilic Esophagitis Endoscopic Reference Score (EREFs) for APT-1011 responders randomized to continue APT-1011 3 mg HS with responders randomized to placebo (withdrawal of APT-1011 3 mg HS). The EREF score has a range from 0-9, with 9 being worst result.
Mean Histologic Change | Week 0 to Week 52
  To compare the mean change from baseline to the end of the RWS in peak eosinophil counts for APT-1011 responders randomized to APT-1011 3 mg HS with those randomized to placebo in the RWS.
Mean Change in PROSE Day-Level Symptom Burden | Week 0 to Week 52
  To compare the mean change in day-level symptom burden using the Patient Reported Outcomes Symptoms of EoE (PROSE) from baseline to the end of RWS, for APT-1011 responders randomized to continue APT-1011 3 mg HS with responders randomized to placebo (withdrawal of APT-1011 3 mg HS). Day-level symptom burden has values ranging from 0 (no symptoms) to 10 (symptoms are as bad as I can imagine).
Mean Change in PROSE Day-Level Difficulty Swallowing | Week 0 to Week 52
  To compare the mean change in day-level difficulty swallowing using the Patient Reported Outcomes Symptoms of EoE (PROSE) from baseline to the end of randomized withdrawal phase, for APT-1011 responders randomized to continue APT-1011 3 mg HS with responders randomized to placebo (withdrawal of APT-1011 3 mg HS). Each symptom is rated on a numeric rating scale (NRS) with values ranging from 0 (not at all) to 10 (as bad as I can imagine).
Mean Change in Dysphagia-Free Days | Week 0 to Week 52
  To compare the mean number of dysphagia-free days from baseline to the end of RWS, for APT-1011 responders randomized to continue APT-1011 3 mg HS with responders randomized to placebo (withdrawal of APT-1011 3 mg HS)
Mean Change in Number of Dysphagia Episodes | Week 0 to Week 52
  To compare mean change in number of dysphagia episodes from baseline at or prior to Week 52 (based on timing of > 6 peak eos/HPF) for APT-1011 responders randomized to continue APT-1011 3 mg HS with those randomized to placebo (withdrawal of APT-1011 3 mg HS)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Dellon, MD, MPH, Principal Investigator — UNC Center for Eosphageal Diseases and Swallowing
Locations (56):
- United States (48):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Gut P.C., dba; Digestive Health Specialists of the Southeast, Dothan, Alabama
  - East View Medical Research, LLC, Mobile, Alabama
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Preferred Research Partners Inc., Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Camarillo Endoscopy Center, Camarillo, California
  - Hope Clinical Research, Canoga Park, California
  - Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - Medical Associates Research Group, San Diego, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Western States Clinical Research Inc., Wheat Ridge, Colorado
  - Western Connecticut Medical Group - Gastroenterology, Danbury, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Encore Borland Groover Clinical Research, Jacksonville, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Summit Clinical Research, Athens, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Michigan Medicine, University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Bozeman Health GI Clinic, Bozeman, Montana
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - University of North Carolina Health Systems (UNC Hospital), Chapel Hill, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Digestive Disease Associates LTD, Wyomissing, Pennsylvania
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - DHAT Research Institute, Garland, Texas
  - Advanced Research Institute, Ogden, Utah
  - Verity Research, Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
- Australia (6):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Swallow Clinic, St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Spain (2):
  - Hosital General de Tomelloso, Tomelloso, Ciudad Real
  - Hospital Universitario Ramón y Cajal (Madrid), Madrid

IPD SHARING:
Plan to Share IPD: No